CLINICAL TRIAL: NCT03696888
Title: Reducing Risky Alcohol Consumption Using Skills-training in the App-form: A Randomized Controlled Study in the General Population.
Brief Title: Skills-training for Reducing Risky Alcohol Use in App Form
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anne H Berman, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016/1088-31
Record Dates: First submitted 2018-10-02; First posted 2018-10-05 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Alcohol Abuse; Alcohol Use Disorder; Alcohol Drinking; Alcohol Dependence; Alcohol; Harmful Use
Keywords: Randomized Controlled Trial; Internet; Mobile phone; Smartphone; App; Alcohol; Substance use
MeSH Terms: conditions — Alcoholism; Alcohol Drinking; Alzheimer Disease; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Note: A pilot period with interim 6-week analyses following recruitment of about 10% of the maximum anticipated sample of 1000 is part of the study. This offers an opportunity to assess trial continuation from an ethical perspective. The rationale for this is that individuals with relatively severe levels of alcohol use can be included in the trial and the investigators harbor a concern that the components in the intervention and control conditions might be insufficient to support the participants in remaining stable or reducing their alcohol intake. The pilot period covers a recruitment period from Dec 7, 2019 to February 15, 2019 (n=89) and includes a 6-week follow-up. The interim analysis from May 1, 2019 indicates group declines in alcohol use over the 6-week follow-up period for both conditions, suggesting that continuation of the trial is warranted. Pilot participants will be included in the final study sample.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telecoach (Experimental): A skills-training web-app teaching skills for reducing problematic alcohol use.
  Interventions: Behavioral: Telecoach
- TeleCoach control (Active Comparator): A web-app giving information on health-related consequences of alcohol consumption.
  Interventions: Behavioral: TeleCoach control

INTERVENTIONS:
Behavioral: Telecoach — A skills-training web-app teaching skills for reducing problematic alcohol use.
  Arms: Telecoach
Behavioral: TeleCoach control — A web-app providing information about the health-related consequences of alcohol consumption.
  Arms: TeleCoach control

SUMMARY:
This study evaluates the efficacy of a skills training web-based mobile phone application, Telecoach among individuals in the general population seeking help for their risky alcohol consumption on the Internet. The design is a two-armed randomized controlled design, and outcomes are measured in terms of changes in excessive alcohol use at follow up 6, 12 and 26 weeks after study initiation and baseline data gathering. The Telecoach web app delivers skills training in the form of exercises commonly used in psychosocial interventions for risky alcohol use. The controll condition is a web app providing information on the effects of alcohol on the consumers' health.

DETAILED DESCRIPTION:
This study evaluates the efficacy of a skills training web-based mobile phone application, Telecoach among individuals in the general population seeking help for their risky alcohol consumption on the Internet. The design is a two-armed randomized controlled design, and outcomes are measured in terms of changes in excessive alcohol use at follow up 6, 12 and 26 weeks after study initiation and baseline data gathering.

Individuals seeking help for problematic alcohol use on the internet will get access to a webpage with information about the study. Individuals leaving informed consent are asked to fill out questionnaires about alcohol use, depression, anxiety and information on gender and weight. Those with excessive alcohol use (>14 standard glasses/week for men and > 9 for women) are randomized into one of two groups: 1. Access to the Telecoach web-app and 2. Access to a control condition with an information-providing web-app.

Outcomes on alcohol use are gathered by electronic self-registration at 6, 12 and 26 weeks after study initiation. Additional questions on the users' satisfaction with the app assigned to them and other support for problematic alcohol used during the research period at 26 weeks.

The Telecoach web-app is a skills-training app developed for use on a mobile smart-phone. The skills-training components are common to psychosocial treatment protocols for problematic alcohol consumption.

The control condition web-app is a simple text-based app providing information on the effects of alcohol on the consumers' health.

Outcomes will be reported, analyzed and discussed in a scientific article.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* Risky alcohol consumption defined as Alcohol Use Disorders Identification Test (AUDIT) scores of ≥6 points for women and ≥ 8 points for men.

Exclusion Criteria:

* Severe depression, defined as a MADRS-S score of > 30
* Sucide risk, defined as a MADRS-S, item 9 (Lust for life) score > 4
* Drug abuse, defined as a score of ≥ 8 on the DUDIT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 678 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Change in alcohol consumption according to the 7-day Timeline Followback (TLFB) | Time between screening measure and 26-week followup
  Change in the total number of standard glasses (12g of ethanol) consumed for each day of the preceding 7 days at each timepoint compared.

SECONDARY OUTCOMES:
Daily Drinking Questionnaire (DDQ) | Baseline, 6, 12 and 26 week followups.
  The number of standard glasses (12g of ethanol) consumed and over how many hours for each day of a typical week the last month.
Alcohol Use Disorders Identification Test (AUDIT) | Baseline and 26-week followup.
  10 questions measuring alcohol consumption and alcohol-related problems.
Change in alcohol consumption according to the 7-day Timeline Followback (TLFB) | Baseline, 6- and 12-week followups.
  Change in the total number of standard glasses (12g of ethanol) consumed for each day of the preceding 7 days at each timepoint compared.
Readiness Ruler | Baseline and 26-week followup.
  A visual analogue scale measuring participants' motivation to change their alcohol consumption.
DSM-5 Alcohol use disorder criteria. | Baseline
  Criteria for the diagnosis Alcohol use disorder in the the 5th edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5)
Penn Alcohol Craving Scale (PACS) | Baseline, 6, 12 and 26 week followups.
  5 items to measure participants' craving for alcohol.
Alcohol Abstinence Self Efficacy scale (AASE) | Baseline, 6, 12 and 26 week followups.
  12 items for measuring self efficacy in the domain of abstaining from drinking alcohol.
Drug Use Disorders Identification Test (DUDIT) | Baseline
  11 items for measuring participants' drug consumption and drug-related problems.
Montgomery Åsberg Depression Rating Scale - Self-rating version (MADRS-S) | Baseline, 6, 12 and 26 week followups.
  9 questions measuring symptoms of depression
Generalized Anxiety Disorder-7 (GAD-7) | Baseline, 6, 12 and 26 week followups.
  7 questions measuring symptoms of anxiety
Treatment questions (7 questions regarding access to other help and support for problematic alcohol use). | Baseline and 26 week followup.
  7 questions regarding access to other help and support for problematic alcohol use.
Usability questions regarding the participants' experience of using the web-app they were assigned. | 26 week followup
  Questions regarding the participants' experience of using the web-app they were assigned.

CONTACTS AND LOCATIONS:
Overall Officials: Anne H Berman, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska institutet, Department of Clinical Neuroscience, Center for Psychiatric Research, Stockholm, Sweden

REFERENCES:
- [Derived] Berman AH, Molander O, Tahir M, Tornblom P, Gajecki M, Sinadinovic K, Andersson C. Reducing Risky Alcohol Use via Smartphone App Skills Training Among Adult Internet Help-Seekers: A Randomized Pilot Trial. Front Psychiatry. 2020 May 27;11:434. doi: 10.3389/fpsyt.2020.00434. eCollection 2020. PMID 32536880